CLINICAL TRIAL: NCT02245217
Title: Multi-Tracer Positron Emission Tomography (PET) Prediction and Assessment of Response to Gemcitabine in Pancreatic Cancer Patients
Brief Title: Multi-Tracer PET Prediction and Assessment of Response to Gemcitabine in Pancreatic Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI74163
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET/CT Imaging arm (Experimental)
  Interventions: Device: PET/CT scan to assess treatment efficacy

INTERVENTIONS:
Device: PET/CT scan to assess treatment efficacy

SUMMARY:
Study of multi-tracer PET scans to assess response to gemcitabine in pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients must have either

  1. histologically/cytologically-confirmed borderline resectable pancreatic cancer and be prescribed neoadjuvant gemcitabine-plus-Abraxane as part of their standard of care
  2. histologically/cytologically-confirmed locally advanced unresectable pancreatic cancer and be prescribed neoadjuvant gemcitabine-plus-Abraxane as part of their standard of care.
* Diagnostic quality abdominal imaging (CT or MRI) within the past 45 days.
* Patients must be 18 years or older for inclusion in this research study. There is little experience with the safety of fluorine-18 (18F) fluorothymidine (FLT) in children and therefore this radiopharmaceutical should not be used in patients under the age of 18.
* Patients must be willing to lie flat on their back in the PET/CT scanner for up to 2 hours to allow the imaging data to be obtained.
* Patients must document their willingness to be followed for up to 24 months following enrollment in this imaging trial. By signing informed consent, the patients will document their agreement to have clinical and radiographic endpoints and the results of histopathologic tissue analysis and other laboratory information entered into a research database.
* All patients must sign a written informed consent and HIPAA authorization in accordance with institutional guidelines.
* Determination of pregnancy status: Female patients who are not postmenopausal or surgically sterile will undergo a serum pregnancy test prior to baseline and the subsequent set of multi-tracer PET scans. The serum pregnancy test must be performed within 48 hours prior to research PET imaging. A negative test will be necessary for such patients to undergo research PET imaging.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Adequate organ function and laboratory parameters as defined laboratory testing.

Exclusion Criteria:

* Any prior systemic or investigational therapy for pancreatic cancer.
* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals (patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion).
* Patients who are pregnant or lactating or who suspect they might be pregnant. - Serum pregnancy tests will be obtained prior to the baseline and subsequent multi-tracer PET scans in female patients that are not postmenopausal or surgically sterile.
* Adult patients who require monitored anesthesia for PET scanning.
* Patients known to be HIV positive. This is due to the potential toxicities of [18F]FLT in HIV positive patients.
* Pre-existing sensory neuropathy greater than grade 1.
* Prior malignancy except for adequately treated basal cell skin cancer, in situ cervical cancer or any other form of cancer from which the patient has been disease-free for 5 years.
* Uncontrolled diabetes or blood glucose greater than 180 mg/dl on the day of the [18F] fluorodeoxyglucose (FDG) PET scan.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Any other condition that would, in the Investigator's judgment, contraindicate patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, social complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PET/CT Imaging Arm: Positron Emission Tomography (PET)/CT scan to assess treatment efficacy
Period: Overall Study
Arm/Group | PET/CT Imaging Arm
Started | 9
Completed | 7
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- PET/CT Imaging Arm: PET/CT scan to assess treatment efficacy
Arm/Group | PET/CT Imaging Arm
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 67 [54 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: FDG Therapeutic Responses to 1 Cycle
Description: The patients underwent baseline and repeat PET/CT imaging (after one cycle) with fluorodeoxyglucose (FDG) and fluorothymidine (FLT). The percent change in the SUVmax for FDG was determined. From these percent change determinations, a response determination was obtained based on the EORTC criteria. EORTC response criteria define a response as >25% reduction in SUVmax.
Time Frame: 1 month
Measure: Number; unit: participant responses based on EORTC
Arm/Group | PET/CT Imaging Arm
Number analyzed (Participants) | 7
participant responses based on EORTC | 6

2. Primary Outcome: FLT Therapeutic Responses to 1 Cycle
Description: The patients underwent baseline and repeat PET/CT imaging (after one cycle) with FDG and FLT. The percent change in the SUVmax for FLT was determined. From these percent change determinations, a response determination was obtained based on the EORTC criteria. EORTC response criteria define a response as >25% reduction in SUVmax.
Time Frame: 1 month
Population: Patients who completed both baseline and follow-up imaging. A synthesis failure for FLT occurred on the follow-up imaging for one patient, so that patient was excluded from the FLT analysis.
Measure: Number; unit: participant responses based on EORTC
Arm/Group | PET/CT Imaging Arm
Number analyzed (Participants) | 6
participant responses based on EORTC | 1

3. Primary Outcome: RECIST 1.1 Therapeutic Responses to 1 Cycle
Description: The patients underwent baseline and repeat PET/CT imaging (after one cycle) with FDG and FLT. Tumor response was determined by RECIST 1.1 and defined as a >30% reduction in tumor size as determined by the sum of the longest diameters of each index lesion
Time Frame: 1 month
Measure: Number; unit: participant responses based on RECIST1.1
Arm/Group | PET/CT Imaging Arm
Number analyzed (Participants) | 7
participant responses based on RECIST1.1 | 3

ADVERSE EVENTS:
Arm/Group | PET/CT Imaging Arm
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes